CLINICAL TRIAL: NCT03746431
Title: A Phase 1 Study of [225Ac]-FPI-1434 Injection in Patients With Locally Advanced or Metastatic Solid Tumours
Brief Title: A Phase 1 Study of [225Ac]-FPI-1434 Injection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A strategic decision was made to discontinue the study and prioritize other programs within the portfolio. The study was not discontinued due to safety issues or adverse events related to FPI-1434, FPE-1547, or FPI-1175.
Sponsor: Fusion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FPX-01-01
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumours; Endometrial Cancer; Cervical Cancer; Ovarian Cancer; Breast Cancer; Triple Negative Breast Cancer (TNBC); HER2-negative Breast Cancer; Head and Neck Squamous Cell Carcinoma (HNSCC); Adrenocortical Carcinoma; Uveal Melanoma
Keywords: 225-Ac Labelled Humanized Monoclonal Antibody Against IGF-1R; [225Ac]-FPI-1434; IGF-IR Targeted Alpha Therapeutic; IGF-IR Radioligand Therapy; Radiopharmaceuticals
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Adrenocortical Carcinoma; Uveal Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- [225Ac]-FPI-1434 Single-Dose Escalation (Experimental)
  Interventions: Drug: [111In]-FPI-1547 Injection; Drug: [225Ac]-FPI-1434 Injection single-dose
- [225Ac]-FPI-1434 Multi-Dose Escalation (Experimental): [225Ac]-FPI-1434 treatment with or without pre-administration of FPI-1175 (cold antibody).
  Interventions: Drug: [111In]-FPI-1547 Injection; Drug: [225Ac]-FPI-1434 Injection multi-dose; Biological: FPI-1175 Infusion
- FPI-1175 Cold Antibody (Experimental)
  Interventions: Drug: [111In]-FPI-1547 Injection; Drug: [225Ac]-FPI-1434 Injection multi-dose; Biological: FPI-1175 Infusion
- [225Ac]-FPI-1434 Multi-Dose (Experimental): Phase 2 Tumour Cohort - Head & Neck Squamous Cell Carcinoma (HNSCC), Endometrial Cancer, Cervical Cancer, Ovarian Cancer, Triple Negative Breast Cancer (TNBC), HER2-negative, Adrenocortical Carcinoma (ACC), Uveal Melanoma, [225Ac]-FPI-1434 treatment with or without pre-administration of FPI-1175 (cold antibody).
  Interventions: Drug: [111In]-FPI-1547 Injection; Drug: [225Ac]-FPI-1434 Injection multi-dose; Biological: FPI-1175 Infusion

INTERVENTIONS:
Drug: [111In]-FPI-1547 Injection — [111In]-FPI-1547 is a targeted radioimmuno-imaging agent that consists of FPI-1175, an insulin-like growth factor-1 receptor (IGF-1R)-targeting humanized monoclonal antibody, a bifunctional chelate, and Indium-111, a radionuclide. Patients will receive [111In]-FPI-1547 Injection of 185 MBq (5 mCi) for imaging.
Drug: [225Ac]-FPI-1434 Injection multi-dose — [225Ac]-FPI-1434 is a targeted alpha radioimmuno-therapeutic agent that consists of FPI-1175, an insulin-like growth factor-1 receptor (IGF-1R)-targeting humanized monoclonal antibody, a bifunctional chelate, and Actinium-225, an alpha-emitting radionuclide. Patients will receive multiple doses of [225Ac]-FPI-1434 Injection. Dose is per cohort assignment.
  Arms: FPI-1175 Cold Antibody; [225Ac]-FPI-1434 Multi-Dose; [225Ac]-FPI-1434 Multi-Dose Escalation
Biological: FPI-1175 Infusion — FPI-1175 is an insulin-like growth factor-1 receptor (IGF-1R)-targeting humanized monoclonal antibody without a radioisotope. Patients will receive FPI-1175 Infusion at a dose per cohort assignment.
  Arms: FPI-1175 Cold Antibody; [225Ac]-FPI-1434 Multi-Dose; [225Ac]-FPI-1434 Multi-Dose Escalation
Drug: [225Ac]-FPI-1434 Injection single-dose — [225Ac]-FPI-1434 is a targeted alpha radioimmuno-therapeutic agent that consists of FPI-1175, an insulin-like growth factor-1 receptor (IGF-1R)-targeting humanized monoclonal antibody, a bifunctional chelate, and Actinium-225, an alpha-emitting radionuclide. Patients will receive a single dose of [225]-FPI-1434 Injection. Dose is per cohort assignment.
  Arms: [225Ac]-FPI-1434 Single-Dose Escalation

SUMMARY:
This is a first-in-human Phase 1/2, non-randomized, multi-centre, open-label clinical study designed to investigate safety, tolerability, PK, and preliminary anti-tumour activity of [225Ac]-FPI-1434 (radioimmuno-therapeutic agent) in patients with solid tumours that demonstrate uptake of [111In]-FPI-1547 (radioimmuno-imaging agent), and to establish the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of repeat doses of [225Ac]-FPI-1434 Injection in patients with solid tumours that demonstrate uptake of [111In]-FPI-1547 (radioimmuno-imaging agent).

DETAILED DESCRIPTION:
This study consists of a Phase 1 portion and a Phase 2 portion.

Phase 1 includes the following cohorts: Single dose-ascending cohorts and Multi- dose ascending cohorts of [225Ac]-FPI-1434 and Multi- dose ascending cohorts evaluating administration of FPI-1175 (cold antibody), followed by, [225Ac]-FPI-1434 (cold + hot), with cycles repeating every 42 days. And Cold Antibody Sub-study evaluating administration of ascending doses of FPI-1175 followed by [111In]-FPI-1547.

The Phase 2 will evaluate [111In]-FPI-1547 and [225Ac]-FPI-1434 with or without FPI-1175 in tumour-specific cohorts. The decision to utilize FPI-1175 in the Phase 2 portion of the study will be determined based on Phase 1 data, including safety, tolerability, pharmacokinetic and dosimetry results.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically documented, definitively diagnosed, advanced solid tumour that is refractory to all standard treatment, for which no standard treatment is available, or it is contraindicated, or the patient refuses standard therapy.
2. Measurable or evaluable disease in accordance with RECIST 1.1.
3. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
4. Life expectancy of greater than 3 months as judged by the treating physician.
5. Available tumour tissue (either archival or fresh biopsy) for IGF-1R immunohistochemistry. Submission of the tissue is not required prior to enrollment.
6. Adequate heart, kidney, and liver function
7. Adequate bone marrow reserves
8. Ability to understand and the willingness to sign a written informed consent document.

   Phase 2 Specific
9. Histologically and/or cytologically documented diagnosis of locally advanced, inoperable, metastatic, or recurrent solid tumour types: endometrial, cervical, ovarian, TNBC, HER 2-negative breast, HNSCC, ACC, or uveal melanoma.
10. Have measurable disease per RECIST 1.1 Failure to respond to standard systemic therapy, or for whom standard or curative systemic therapy does not exist or is not tolerable.

    Imaging Eligibility
11. Prior to the initial [225Ac]-FPI-1434 cycle: Sufficient target expression in at least 1 lesion following [111In]-FPI-1547 and SPECT imaging.

Exclusion Criteria:

1. Systemic therapeutic radiopharmaceutical within 6 months prior to enrollment into this study.
2. Contraindications to or inability to perform the required imaging procedures in this study (e.g., inability to lay flat during scan time)
3. Uncontrolled brain metastasis, including but not limited to the need for treatment with steroids, surgery or radiation therapy.
4. Anticancer therapy (including investigational agents) or external beam radiation therapy within 14 days of the dosing of [111In]-FPI-1547
5. Has known additional malignancy that is progressing or has required active treatment within the past 3 years. Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast cancer, cervical cancer, prostate) that have undergone potentially curative therapy are not excluded.
6. Residual CTCAE ≥ Grade 2 side effects of prior therapy, with the exception of residual grade 2 alopecia.
7. Prior organ transplantation, including stem cell transplantation.
8. Any prior treatment with nitrosoureas or actinomycin-D.
9. Clinically relevant levels of protein in the urine
10. Known or suspected allergies or contraindications to the Investigational Products or any component of the investigational drug formulation.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Received > 20 Gy prior radiation to large areas of the bone marrow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Incidence of adverse events (AEs). | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1
Single-Dose Escalation: Incidence of dose limiting toxicities (DLTs). | 8 weeks.
  Phase 1
Multi-Dose Escalation: Incidence of DLTs. | 6 weeks.
  Phase 1
Dose Escalation: Incidence of clinically significant clinical laboratory abnormalities. | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1
Dose Escalation: Changes in electrocardiogram (ECG) parameters (PR, QRS, QT, and QTc intervals). | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1
Cold Antibody Sub-Study: Changes in uptake of [111In]-FPI-1547 Injection following FPI-1175 Infusion in selected regions of interest on SPECT/CT images. | Within two weeks of the first [111In]-FPI-1547 Injection.
  Phase 1
Cold Antibody Sub-Study: Changes in radiation dose estimates for selected tissues, organs and whole body both for [111In]-FPI-1547 and [225Ac]-FPI-1434 Injection at various dose levels following FPI-1175 Infusion. | Within two weeks of the first [111In]-FPI-1547 Injection.
  Phase 1
Evaluate anti-tumour activity of [225Ac]-FPI-1434 regimen | Approximately one year post final [225Ac]-FPI-1434 injection.
  Phase 2
Objective response rate (ORR) RECIST v1.1. | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 2

SECONDARY OUTCOMES:
Dose Escalation and Cold Antibody Sub-Study: Tumour uptake of [111In]-FPI-1547 in selected regions of interest on SPECT/CT images. | Dose Escalation: Within one week of the [111In]-FPI-1547 Injection. Cold-Antibody Sub-Study: Within two weeks of the first [111In]-FPI-1547 Injection.
  Phase 1 and 2
Dose Escalation: Radiation doses for selected organs and whole body both for [111In]-FPI-1547 Injection and [225Ac]-FPI-1434 Injection. | Within one week of the [111In]-FPI-1547 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Changes in radiation absorbed doses for tumour lesions for [225Ac]-FPI-1434. | Dose Escalation: Within one week of the [111In]-FPI-1547 Injection. Cold-Antibody Sub-Study: Within two weeks of the first [111In]-FPI-1547 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Clearance for radioactivity and for the targeting antibody. | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Area under the curve (AUC) for radioactivity and for the targeting antibody. | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Cmax for radioactivity and for the targeting antibody. | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Half-life for radioactivity and for the targeting antibody. | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Objective response rate (ORR) (sum of complete and partial response) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Prostate Cancer Working Group 3 (PCWG3) guidelines. | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1
Dose Escalation: Changes in the corrected QT (QTc) interval in milliseconds after [225Ac]-FPI-1434 treatment, compared to baseline. | Approximately 24 hours from the time of [225Ac]-FPI-1434 Injection administration.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Changes in human growth hormone (hGh) following [111In]-FPI-1547 Injection and [225Ac]-FPI-1434 Injection. | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Changes in insulin-like growth factor 1 (IGF-1) following [111In]-FPI-1547 Injection and [225Ac]-FPI-1434 Injection. | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Changes in insulin-like growth factor binding protein 3 (IGFBP-3) following [111In]-FPI-1547 Injection and [225Ac]-FPI-1434 Injection. | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Cold Antibody Sub-Study: Incidence of AEs. | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Cold Antibody Sub-Study: Incidence of clinically significant clinical laboratory abnormalities. | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Cold Antibody Sub-Study: Changes in ECG parameters (PR, QRS, QT, and QTc intervals). | 4 weeks post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Time to response (TTR). | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Duration of response (DoR). | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Progression free survival (PFS). | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Time to Progression (TTP). | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Disease control rate (DCR). | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2
Dose Escalation and Cold-Antibody Sub-Study: Overall survival (OS). | Approximately one year post final [225Ac]-FPI-1434 Injection.
  Phase 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Julia Kazakin, MD, Study Director — Fusion Pharmaceuticals Inc.
Locations (13):
- United States (7):
  - City of Hope, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Heidelberg, Victoria
- Canada (4):
  - Juravinski Cancer Center - Hamilton Health, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier De I'Universite de Montreal, Montreal, Quebec
  - Quebec University Hospital- Laval, Québec, Quebec

REFERENCES:
- [Derived] Anderson PM, Subbiah V, Trucco MM. Current and future targeted alpha particle therapies for osteosarcoma: Radium-223, actinium-225, and thorium-227. Front Med (Lausanne). 2022 Nov 15;9:1030094. doi: 10.3389/fmed.2022.1030094. eCollection 2022. PMID 36457575
- [Derived] Martiniova L, Zielinski RJ, Lin M, DePalatis L, Ravizzini GC. The Role of Radiolabeled Monoclonal Antibodies in Cancer Imaging and ADC Treatment. Cancer J. 2022 Nov-Dec 01;28(6):446-453. doi: 10.1097/PPO.0000000000000625. PMID 36383907